CLINICAL TRIAL: NCT04088188
Title: A Phase I, Multi-Center, Open Label, Dose De-Escalation and Expansion Study of Gemcitabine and Cisplatin With AG120 or Pemigatinib for Advanced Cholangiocarcinoma
Brief Title: Gemcitabine and Cisplatin With Ivosidenib or Pemigatinib for the Treatment of Unresectable or Metastatic Cholangiocarcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-ICRN-1701; NCI-2019-05811 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-ICRN-1701 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-04

CONDITIONS: Advanced Cholangiocarcinoma; Metastatic Cholangiocarcinoma; Unresectable Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine; ivosidenib; pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (ivosidenib, cisplatin, gemcitabine) (Experimental): Patients receive ivosidenib PO on days 1-21, cisplatin IV on days 1 and 8, and gemcitabine IV on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Ivosidenib
- Arm B (pemigatinib, cisplatin, gemcitabine) (Experimental): Patients receive pemigatinib PO on days 1-21, cisplatin IV on days 1 and 8, and gemcitabine IV on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Pemigatinib

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Drug: Ivosidenib — Given PO
  Other Names: AG-120; Tibsovo
  Arms: Arm A (ivosidenib, cisplatin, gemcitabine)
Drug: Pemigatinib — Given PO
  Other Names: INCB054828; Pemazyre
  Arms: Arm B (pemigatinib, cisplatin, gemcitabine)

SUMMARY:
This phase I trial studies the side effects and best dose of gemcitabine and cisplatin when given together with ivosidenib or pemigatinib in treating patients with cholangiocarcinoma that cannot be removed with surgery (unresectable) or has spread to other places in the body (metastatic). Chemotherapy drugs, such as gemcitabine and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Ivosidenib and pemigatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving gemcitabine and cisplatin with ivosidenib or pemigatinib may work better in treating patients with cholangiocarcinoma compared to gemcitabine and cisplatin alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety, tolerability, maximum tolerated dose (MTD) and/or recommended phase 2 dose, gemcitabine and cisplatin in combination with either ivosidenib or pemigatinib.

SECONDARY OBJECTIVES:

I. To evaluate median and progression free survival (PFS) for 6 months per investigator assessment.

II. To evaluate the rate of overall survival (OS) in patients treated with gemcitabine and cisplatin in combination with either ivosidenib or pemigatinib.

III. To describe the overall toxicity and adverse events profile associated with gemcitabine and cisplatin in combination with either ivosidenib or pemigatinib.

IV. To determine the best response profile per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria in patients treated with gemcitabine and cisplatin in combination with either ivosidenib or pemigatinib.

CORRELATIVE RESEARCH OBJECTIVE:

I. To measure plasma 2-hydroxglutarate (2-HG) levels =< 21 days prior to registration and at cycle 4 day 1 (+/- 2 days).

OUTLINE: This is a dose de-escalation study. Patients are assigned to 1 of 2 arms.

ARM A (IDH1 GENE MUTATION): Patients receive ivosidenib orally (PO) on days 1-21, cisplatin intravenously (IV) on days 1 and 8, and gemcitabine IV on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM B (FGFR2 GENE ALTERATION): Patients receive pemigatinib PO on days 1-21, cisplatin IV on days 1 and 8, and gemcitabine IV on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis (fresh) or banked tumor biopsy sample collected within the last 3 years from the registration date consistent with nonresectable or metastatic cholangiocarcinoma and are not eligible for curative resection, transplantation, or ablative therapies
* Documented disease without any evidence of progression following at least 3 cycles of standard-of-care chemotherapy including gemcitabine and cisplatin as part of first-line systemic therapy; NOTE: Only patients receiving standard-of-care chemotherapy including gemcitabine and cisplatin as first-line therapy for unresectable or metastatic cholangiocarcinoma will be permitted to enroll in this trial. Prior systemic adjuvant chemotherapy is allowed as long as there was no evidence of recurrence within 6 months of completing the adjuvant therapy
* Molecular testing result from Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory (using fresh tumor biopsy or most recent banked tumor tissue available) confirming that the tumor tissue has at least one of the following:

  * IDH1 gene mutation (R132C/L/G/H/S mutation)
  * FGFR2 gene alteration
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Life expectancy >= 3 months
* At least one evaluable and measurable lesion by RECIST criteria prior to beginning chemotherapy with gemcitabine and cisplatin

  * NOTE: Subjects who have received prior local therapy (including but not limited to embolization, chemoembolization, radiofrequency ablation, hepatic arterial infusion, or radiation therapy) are eligible provided measurable disease falls outside of the treatment
* Recovered from toxicities associated with prior anticancer therapy to baseline unless stabilized under medical management
* Absolute neutrophil count >= 1,500/mm^3 (obtained =< 21 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 21 days prior to registration)
* Hemoglobin >= 8 g/dL (obtained =< 21 days prior to registration)
* Serum total bilirubin =< 2.0 x upper limit of normal (ULN), unless considered due to Gilbert's disease. If Gilbert's disease or disease involving liver, serum total bilirubin =< 2.5 x ULN (obtained =< 21 days prior to registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN or =< 5.0 x ULN in the presence of liver metastases (obtained =< 21 days prior to registration)
* Serum creatinine < 1.5 x ULN OR creatinine clearance >= 50 mL/min based on the Cockcroft-Gault glomerular filtration rate (GFR) estimation (obtained =< 21 days prior to registration)
* Serum phosphate =< institutional ULN and potassium within institutional normal range for Arm B only (obtained =< 21 days prior to registration)

  * NOTE: Supplemental potassium may be used to correct potassium prior to registration
* Negative serum pregnancy test done =< 7 days prior to registration for women of childbearing potential only

  * NOTE: Females of reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy, or tubal occlusion or who have not been naturally postmenopausal (i.e., who have not menstruated) for >= 24 consecutive months (i.e., have not had menses at any time in the preceding 24 consecutive months)
* Women of reproductive potential and fertile men must agree to use 2 effective forms of contraception (including at least 1 barrier form) from the time of giving informed consent throughout the study and for 90 days (both females and males) following the last dose of study drug

  * NOTE: Effective forms of contraception are defined as hormonal oral contraceptives, injectables, patches, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal ligation, condoms with spermicide, or male partner sterilization
* Able to understand and willing to sign the informed consent form

  * NOTE: A legally authorized representative may consent on behalf of a subject who is otherwise unable to provide informed consent if acceptable to and approved by the site's Institutional Review Board (IRB)/Independent Ethics Committee (IEC)
* Able to comply with scheduled visits, treatment plans, procedures, and laboratory tests, including serial peripheral blood sampling during the study
* Willing to provide blood samples for correlative research purposes

Exclusion Criteria:

* Prior therapy with either an IDH inhibitor or selective FGFR inhibitor

  * IDH inhibitors: ivosidenib, FT-2012, etc.
  * FGFR inhibitors: pemigatinib, BGJ-398, TAS-120, ARQ 087, or derazantinib, etc.
* Progressive disease as best response on current standard-of-care chemotherapy including gemcitabine and cisplatin
* Known toxicity to standard-of-care chemotherapy including gemcitabine and cisplatin requiring cessation of this therapy
* Received radiotherapy to metastatic sites of disease =< 2 weeks prior to registration
* Underwent hepatic radiation, chemoembolization, or radiofrequency ablation =< 4 weeks prior to registration
* Known symptomatic brain metastases requiring steroids

  * NOTE: Subjects with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study entry, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and have radiographically stable disease for at least 3 months prior to registration
  * NOTE: Up to 10 mg per day of prednisone equivalent will be allowed
* Other active malignancy =< 5 years prior to registration. EXCEPTIONS:

  * Non- melanoma skin cancer unless stage 1a or carcinoma-in-situ of the cervix
  * Breast cancer with ongoing hormone therapy being administered as adjuvant therapy

    * NOTE: If there is a history or prior malignancy, they must not be receiving other specific treatment
* Major surgery =< 4 weeks prior to registration or have not recovered from post-surgery toxicities
* Any of the following because this study involves investigational agents whose genotoxic, mutagenic, and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Arm A: Use of strong CYP3A4 inducers or strong or moderate CYP3A4 inhibitors. In addition, sensitive CYP3A4 substrate medications with a narrow therapeutic window, unless they can be transferred to other medications =< 4 days or 5 half-lives (whichever is shorter) prior to registration
* Arm B: Use of strong CYP3A4 inducers or inhibitors or moderate CYP3A4 inducers
* NOTE: Study principal investigator (PI) approval is needed if continued use of CYP3A4 inducers or inhibitors. Approval can be obtained via email (documentation of approval/eligibility needed)
* For Arm B only: Current evidence of clinically significant corneal (including but not limited to bullous/band keratopathy, corneal abrasion, inflammation/ulceration, and keratoconjunctivitis) or retinal disorder (including but not limited to central serous retinopathy, macular/retinal degeneration, diabetic retinopathy, retinal detachment) as confirmed by ophthalmologic examination
* Known history and/or current evidence of ectopic mineralization/ calcification, including but not limited to soft tissue, kidneys, intestine, myocardia, or lung, excepting calcified lymph nodes and asymptomatic arterial or cartilage/tendon calcification for Arm B only
* Known history of hypovitaminosis D requiring supraphysiologic doses to replenish the deficiency for Arm B only

  * NOTE: Subjects receiving vitamin D food supplements are allowed
* Active infection requiring systemic anti-infective therapy or with an unexplained fever > 38.5 degrees Celsius (C) =< 7 days of registration

  * NOTE: At the discretion of the investigator, subjects with tumor fever may be enrolled
* Any known hypersensitivity to any of the components of ivosidenib or pemigatinib
* Significant, active cardiac disease =< 6 months prior to registration, including

  * New York Heart Association (NYHA) class III or IV congestive heart failure
  * Myocardial infarction
  * Unstable angina
  * Stroke
* Have a heart-rate corrected QT interval (using Fridericia's formula) (QTcF) >= 450 msec or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome)

  * Note: Bundle branch block and prolonged QTcF interval are permitted with approval of the medical monitor
* Taking medications that are known to prolong the QT interval, unless they can be transferred to other medications >= 5 half-lives prior to registration or unless the medications can be properly monitored during the study

  * Note: If equivalent medication is not available, QTcF should be closely monitored
* Known active hepatitis B (hepatitis B virus [HBV]) or hepatitis C (hepatitis C virus [HCV]) infections, known positive human immunodeficiency virus (HIV) antibody results, or acquired immunodeficiency syndrome (AIDS) related illness

  * NOTE: Subjects with a sustained viral response to HCV or immunity to prior HBV infection will be permitted. Subjects with chronic HBV that is adequately suppressed per institutional practice will be permitted
  * NOTE: HBV, HCV, and/or HIV testing is not required prior to trial registration
* Any other acute or chronic medical or psychiatric condition, including recent (=< 12 months of registration) or active suicidal ideation or behavior, or a laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study
* Inability or unwillingness to swallow ivosidenib or pemigatinib or have significant gastrointestinal (GI) disorder(s) that could interfere with absorption, metabolism, or excretion

  * NOTE: Gastroesophageal reflux disease under medical treatment is allowed (assuming no drug interaction potential)
* Have been committed to an institution by virtue of an order issued either by the judicial or administrative authorities
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shubham Pant, Principal Investigator — Academic and Community Cancer Research United
Locations (7):
- United States (7):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Spartanburg Regional Medical Center, Forest City, North Carolina
  - M D Anderson Cancer Center, Houston, Texas
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Ivosidenib, Cisplatin, Gemcitabine): Patients receive ivosidenib PO at a starting dose of 500mg on days 1-21, cisplatin IV on days 1 and 8, and gemcitabine IV on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Arm B (Pemigatinib, Cisplatin, Gemcitabine): Patients receive pemigatinib PO at a starting dose of 13.5mg on days 1-21, cisplatin IV on days 1 and 8, and gemcitabine IV on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A (Ivosidenib, Cisplatin, Gemcitabine) | Arm B (Pemigatinib, Cisplatin, Gemcitabine)
Started | 6 | 1
Completed | 2 | 1
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: Arms A and B are reported together to maintain patient deidentification and privacy.
Groups:
- Arm A (Ivosidenib, Cisplatin, Gemcitabine) and Arm B (Pemigatinib, Cisplatin, Gemcitabine): Arm A patients receive ivosidenib PO at a starting dose of 500mg on days 1-21, cisplatin IV on days 1 and 8, and gemcitabine IV on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Arm B patients receive pemigatinib PO at a starting dose of 13.5mg on days 1-21, cisplatin IV on days 1 and 8, and gemcitabine IV on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm A (Ivosidenib, Cisplatin, Gemcitabine) and Arm B (Pemigatinib, Cisplatin, Gemcitabine)
Number analyzed (Participants) | 7
Age, Continuous [Mean (Full Range); unit: years] | 54.7 [29 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Primary Tumor Site [Count of Participants; unit: Participants]
  Extrahepatic bile duct | 1
  Intrahepatic bile ducts | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Significant Toxicities
Description: A significant toxicity is defined as a Dose Limiting Toxicity that is possibly, probably, or definitely related to treatment. DLTs will be evaluated starting in the first cycle of combination treatment and up to 3 weeks of combination treatment. Toxicities will be assessed using the CTEP Active Version of the CTCAE. All patients meeting the eligibility criteria who have signed a consent form and have begun combination treatment will be considered evaluable for significant toxicity. Patients, who do not experience a DLT but withdraw from protocol therapy prior to 3 weeks, will not be evaluable for the primary endpoint. Incidence of significant toxicity at 3 weeks will be estimated separately by arm and will be defined as the number of patients with significant toxicity within 3 weeks of combination treatment divided by the total number of evaluable patients.
Time Frame: 3 weeks
Population: Only patients that completed cycle 1 treatment per protocol were evaluated.
Measure: Count of Participants; unit: Participants
Groups:
- Arm B (Pemigatinib, Gemcitabine, Cisplatin): Patients receive pemigatinib PO at a starting dose of 13.5mg on days 1-21, cisplatin IV on days 1 and 8, and gemcitabine IV on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm A (Ivosidenib, Cisplatin, Gemcitabine) | Arm B (Pemigatinib, Gemcitabine, Cisplatin)
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined to be the length of time from start of study therapy to death due to any cause. All patients meeting the eligibility criteria that have signed a consent form and begun treatment will be considered evaluable for estimation of the survival distribution. The distribution of overall survival for both arms of the study will be estimated separately using the Kaplan-Meier method.
Time Frame: 27 months
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- B (Pemigatinib, Cisplatin, Gemcitabine): Patients receive pemigatinib PO at a starting dose of 13.5mg on days 1-21, cisplatin IV on days 1 and 8, and gemcitabine IV on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm A (Ivosidenib, Cisplatin, Gemcitabine) | B (Pemigatinib, Cisplatin, Gemcitabine)
Number analyzed (Participants) | 6 | 1
Months | 22.9 [18.2 to NA] — Upper CI was not met due to a lack of events. | NA [NA to NA] — The median and CI were not able to be computed due to a lack of events.

3. Secondary Outcome: Progression Free Survival
Description: Progression free survival time is defined as the time from the start of study therapy to documentation of disease progression. Patients who die without documentation of progression will be considered to have had tumor progression at the time of death. Patients who are still alive and have not progressed will be censored for progression at the time of the last disease evaluation. The time-to-progression distribution will be estimated separately for both arms, using the Kaplan-Meier method.
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Ivosidenib, Cisplatin, Gemcitabine) | Arm B (Pemigatinib, Cisplatin, Gemcitabine)
Number analyzed (Participants) | 6 | 1
Months | 15.4 [13.8 to NA] — Upper CI was not reached due to a lack of events. | 4.9 [NA to NA] — The CI was unable to be estimated due to a lack of events.

4. Secondary Outcome: Number of Patients Experiencing Adverse Events
Description: The number and severity of all adverse events (overall, by dose-level, and by tumor group) will be tabulated and summarized in this patient population. The grade 3+ adverse events will also be described and summarized in a similar fashion.
Time Frame: 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Ivosidenib, Cisplatin, Gemcitabine) | Arm B (Pemigatinib, Cisplatin, Gemcitabine)
Number analyzed (Participants) | 6 | 1
Participants | 5 | 1

5. Secondary Outcome: Number of Participants Experiencing Toxicities
Description: The term toxicity is defined as adverse events that are classified as either possibly, probably, or definitely related to study treatment. Non-hematologic toxicities will be evaluated via the ordinal Common Terminology Criteria (CTC) standard toxicity grading. Hematologic toxicity measures of thrombocytopenia, neutropenia, and leukopenia will be assessed using continuous variables as the outcome measures (primarily nadir) as well as categorization via CTC standard toxicity grading. Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Time Frame: 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Ivosidenib, Cisplatin, Gemcitabine) | Arm B (Pemigatinib, Cisplatin, Gemcitabine)
Number analyzed (Participants) | 6 | 1
Participants | 4 | 1

6. Secondary Outcome: Best Response
Description: Best Response is defined to be the best objective status recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria. Response Evaluation Criteria in Solid Tumors 1.1 criteria will be used for tumor evaluation and patients will be re-evaluated every prior to treatment in cycle 3 and then in odd subsequent cycles. Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall and by tumor group).
Time Frame: 15 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Ivosidenib, Cisplatin, Gemcitabine) | Arm B (Pemigatinib, Cisplatin, Gemcitabine)
Number analyzed (Participants) | 6 | 1
Participants
  PR | 1 | 0
  SD | 5 | 1

ADVERSE EVENTS:
Time Frame: 27 months
Groups:
- Arm A (Ivosidenib, Cisplatin, Gemcitabine): Arm A patients receive ivosidenib PO at a starting dose of 500mg on days 1-21, cisplatin IV on days 1 and 8, and gemcitabine IV on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Arm B (Pemigatinib, Cisplatin, Gemcitabine): Arm B patients receive pemigatinib PO at a starting dose of 13.5mg on days 1-21, cisplatin IV on days 1 and 8, and gemcitabine IV on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm A (Ivosidenib, Cisplatin, Gemcitabine) | Arm B (Pemigatinib, Cisplatin, Gemcitabine)
All-Cause Mortality (participants affected / at risk) | 3/6 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/1
Other Adverse Events (participants affected / at risk) | 6/6 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Ivosidenib, Cisplatin, Gemcitabine) (N=6) | Arm B (Pemigatinib, Cisplatin, Gemcitabine) (N=1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Ivosidenib, Cisplatin, Gemcitabine) (N=6) | Arm B (Pemigatinib, Cisplatin, Gemcitabine) (N=1)
Anemia (Blood and lymphatic system disorders) | 5 (65) | 1 (4)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (4)
Dry eye (Eye disorders) | 0 (0) | 1 (4)
Eye pain (Eye disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (5) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (4)
Mucositis oral (Gastrointestinal disorders) | 2 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (25) | 1 (3)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0)
Edema face (General disorders) | 1 (2) | 0 (0)
Edema limbs (General disorders) | 1 (3) | 1 (3)
Fatigue (General disorders) | 6 (53) | 1 (4)
Fever (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (2)
Alkaline phosphatase increased (Investigations) | 4 (20) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Creatinine increased (Investigations) | 2 (6) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (7) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (20) | 1 (2)
Platelet count decreased (Investigations) | 5 (34) | 1 (3)
White blood cell decreased (Investigations) | 4 (21) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (10) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (6) | 1 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (8) | 1 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (31) | 0 (0)
Confusion (Psychiatric disorders) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (8) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (12) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (17) | 1 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4)
Flushing (Vascular disorders) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT04088188/Prot_SAP_000.pdf